CLINICAL TRIAL: NCT02806388
Title: Individualized Molecular Profiling for Allocation to Clinical Trials (IMPACT) Project
Acronym: IMPACT
Status: Recruiting | Type: Observational
Sponsor: National Cancer Centre, Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: ECRU-IMPACT
Record Dates: First submitted 2016-06-16; First posted 2016-06-20 (Estimated); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Solid Tumor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Remaining tumor and/or blood and/or saliva and/or pleural fluid and/or FNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- tumor tissue for molecular profiling

SUMMARY:
This study aims to screen tumor molecular profile for better selection of anticancer treatment, in particular, allocation to clinical trials if available.

DETAILED DESCRIPTION:
Molecular profiling will be performed on archival tumor tissue or freshly collected tumor tissue from re-biopsy. Blood, pleural fluid, FNA, and/or saliva may be collected to study the genetic makeup and also to compare the tumor molecular profile. Personalized therapy will be given based on molecular profile.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed histological diagnosis of solid tumor
* Suitable for systematic treatment and clinical trials
* ECOG (Eastern cooperative oncology group) performance status < 2
* Able to provide tumor tissue for molecular profiling
* Able to understand and sign the informed consent form

Exclusion Criteria:

* None

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any advanced cancer patient who would benefit from molecular profiling and is a potential clinical trial candidate as identified by treating physician.
Sampling Method: Probability Sample
Enrollment: 5500 (Estimated)
Dates: Start 2011-10; Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The molecular and clinical epidemiology for cancer patients being considered for novel therapeutics | 5 years

SECONDARY OUTCOMES:
The proportion of patients who have actionable alterations and enrol into clinical trials | 5 years
The correlation of molecular profiles with clinical outcomes | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Daniel SW Tan, Principal Investigator — National Cancer Centre, Singapore
Locations (1):
- National Cancer Centre, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chia S, Low JL, Zhang X, Kwang XL, Chong FT, Sharma A, Bertrand D, Toh SY, Leong HS, Thangavelu MT, Hwang JSG, Lim KH, Skanthakumar T, Tan HK, Su Y, Hui Choo S, Hentze H, Tan IBH, Lezhava A, Tan P, Tan DSW, Periyasamy G, Koh JLY, Gopalakrishna Iyer N, DasGupta R. Phenotype-driven precision oncology as a guide for clinical decisions one patient at a time. Nat Commun. 2017 Sep 5;8(1):435. doi: 10.1038/s41467-017-00451-5. PMID 28874669